CLINICAL TRIAL: NCT01657630
Title: Evaluation of the Use of the Accu-Chek Combo System in Young Patients With Type 1 Diabetes
Brief Title: Accu-Chek Combo in Young Patients
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: Accu-Chek Combo
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Pump Therapy; Type 1 Diabetes; Treatment Satisfaction
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Accu-Chek Combo: 15 type 1 young patients under 6 years old who begin to use the Accu-Chek Combo System
  Interventions: Device: Accu-Chek Combo System

INTERVENTIONS:
Device: Accu-Chek Combo System — 12 weeks using the Accu Chek Combo System, which is an insulin pump system that offers a remote control integrating a bolus calculator, a blood glucose meter, data storage and analysis function.

SUMMARY:
This is an open, prospective, descriptive study aiming to evaluate the change in treatment satisfaction of primary care givers of young children who use the Accu-Chek Combo System. Patients will routinely be scheduled and start their therapy with the Accu-Chek Combo System on visit 1. Twelve weeks later the final acquisition of data will occur. Diabetes Treatment Satisfaction Questionnaires (DTSQ) will be completed at baseline and after 12 weeks, a distinct acceptance questionnaires will be completed at final visit. In addition, Diabetes related therapeutic information will be collected and data about the use of the device components will be downloaded from the Accu-Chek Combo System

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus type 1
* Continuous Subcutaneous Insulin Infusion(CSII)therapy(for at least 6 months)
* Age below 6 years
* Planned and scheduled change to a Accu-Chek Combo System within the next 3 weeks at least
* Signing on an Inform Consent Form

Exclusion Criteria:

* Patient has been diagnosed with progressive/serious diseases that in judgment of the physician preclude successful completion of the observational period
* primary care giver not skilled enough to comment in a qualitative way

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young patients with type 1 Diabetes treated at the institute of Endocrinology and Diabetes, Schneider Children's Medical Center, which is a tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Diabetes Treatment Satisfaction | after 12 weeks
  we will assess patient's treatment satisfaction using Treatment Satisfaction Questionnaires
Study device acceptance | after 12 weeks
  We will assess study device acceptance using a distinct Acceptance Questionnaire

SECONDARY OUTCOMES:
Mean Blood Glucose level | after 12 weeks
  we will compare mean blood glucose level at baseline and after 12 weeks
Number of Hypoglycemia Events | after 12 weeks
  we will compare the number of hypoglycemia events at baseline and after 12 weeks
Number of Hyperglycemia Events | after 12 weeks
  We will compare the number of hyperglycemia events at baseline and after 12 weeks
HbA1c | after 12 weeks
  We will compare HbA1c level at baseline and after 12 weeks
postprandial SMBG (self monitoring blood glucose) | after 12 weeks
  We will compare between postprandial SMBG at baseline and after 12 weeks
Overall number of BG (Blood glucose) measurements | after 12 weeks
  We will compare between number of BG measurements at baseline and after 12 weeks
Number of ketosis events | after 12 weeks
  We will compare number of ketosis events (without documented acidosis with home/hospital management)at baseline and after 12 weeks
Number of Diabetic Ketoacidosis (DKA) events | after 12 weeks
  We will compare number of Diabetic ketoacidosis events at baseline and after 12 weeks
preprandial SMBG (self monitoring blood glucose) | after 12 weeks
  We will compare between preprandial SMBG at baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel